CLINICAL TRIAL: NCT06660238
Title: Assessment of Cerebral Metabolism, Cerebral Blood Flow and Cerebral Oxygen Damage in Patients With Cardiac Arrest Using PET-CT
Brief Title: PET-CT to Assess Brain Damage in Cardiac Arrest Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Tang Ziren, Professor, Capital Medical University
Other Study IDs: 2024-9-26-836
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest; Brain Injuries
Keywords: Cardiac arrest; Positron Emission Tomography-Computed Tomography; cerebral metabolism; cerebral blood flow; cerebral oxygenation
MeSH Terms: conditions — Heart Arrest; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
This was a single-center, observational study. Patients with successful cardiopulmonary resuscitation (CPR) will be transferred to the emergency intensive care unit for further standardized management. After successful return of spontaneous circulation (ROSC) for 72 hours and hemodynamic stability for 24 hours, the patients underwent positron emission computed tomography (PET-CT) examination after resuscitation. The supervising physician accompanied the patient and used monitors to monitor vital signs during the examination. Patients who were on ventilators were mechanically ventilated with a magnetic ventilator (HAMILTON-MRI, United States). In addition to conventional cerebral oxygen metabolism, cerebral blood flow, oxygen extraction fraction, cerebral blood volume and other indicators were added in this experiment. These indicators can evaluate the patient's cerebral metabolism, cerebral blood flow and cerebral blood oxygen damage degree. The neurological outcome was followed up 6 months after onset according to the cerebral performance category（CPC）.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years.
* sustained hemodynamic stability for ≥24h.
* the patients were unconscious and not able to obey verbal commands. • Advanced life support and target temperature management within 6 hours of return of spontaneous circulation (ROSC).

Exclusion Criteria:

* Patients with hemodynamic instability.
* Patients who could not complete cranial PET-CT examination for special reasons. • Patients during pregnancy.
* Patients who combined traumatic brain injury, stroke, cerebral hemorrhage and other diseases.
* Patients whose family members did not agree to be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after successful cardiopulmonary resuscitation (CPR) were transferred to the emergency intensive care unit for further standardized management.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurologic prognosis | 6 months
  Patients will be followed up for neurologic prognosis according to the Cerebral Performance Category Scale（CPC）at 6 months after disease onset.The CPC score was divided into five grades. Grade 1 represented intact brain function, the patient was awake and alert, and had the ability to live and work normally. Grade 2 represents moderate cerebral disability, in which the person is awake and able to work part of the time in a specific environment or perform daily activities independently; Grade 3, severe cerebral disability: the person is awake but dependent on others for daily assistance and retains limited cognition; Grade 4 represents coma and vegetative state, the patient is unconscious, unconscious to the environment, and has no cognitive ability; Level 5 represents death, with the patient confirmed as brain death or death by traditional criteria. According to the CPC score, grade 1-2 was defined as good neurological outcome, and grade 3-5 was defined as poor neurological outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing chaoyang hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: The de-identified survey data will be made available for research purposes by contacting the corresponding authors